CLINICAL TRIAL: NCT02781766
Title: Thrombin Generation Capacity of Patients With Severe Haemophilia Receiving Prophylaxis
Brief Title: TGA (Thrombin Generation Assay) and Prophylaxis in Haemophilia
Acronym: HOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-765
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Haemophilia A
Keywords: Haemophilia A; prophylaxis; thrombin generation assay; factor VIII; prophylactic therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- One arm: patients with severe haemophilia A on prophylaxis (Other): Patients with severe haemophilia A (FVIII < 1 IU/dl), currently on prophylactic therapy , having the same prophylaxis regimen in the last six months, aged between 2 (with a body weight ≥12.5 kg ) and 45 years , with adequate venous access, having patient's diary or equivalent regularly completed and able to give informed consent
  Interventions: Other: Thrombin generation measurement.

INTERVENTIONS:
Other: Thrombin generation measurement.

SUMMARY:
Haemophilic arthropathy is one of the major complications of severe haemophilia. In order to maintain plasma clotting factor activity levels above 1% and avoid spontaneous joint bleeds and other serious bleeding events, prophylactic factor replacement therapy is used. Because of the high cost and limited availability of clotting factor concentrates, dosing is a crucial issue for prophylaxis therapy. Several studies reported a better correlation between clinical bleeding tendency of patients with haemophilia and thrombin generation assay results compared to FVIII/FIX levels. However there is no specific data showing that thrombin generation may be a better indicator of the clinical efficacy of prophylaxis compared to the conventional FVIII measurement.

The main objective of this open, multicentre, prospective study is to compare trough thrombin generation capacity and FVIII levels in severe haemophilia patients and compare these two laboratory results with:

* the number of spontaneous haemarthroses and other spontaneous serious bleeds occurred in the last 6 months
* the number of additional FVIII units used in the last 6 months

This project requires no change in term of type of treatment : During the study, each patient will be treated by his usual clotting factor at the usual regimen (frequency and dosage).

The clinical outcome with the usual prophylaxis regimen will be correlated to TGA results

ELIGIBILITY:
Inclusion Criteria:

* Severe haemophilia A (FVIII < 1 IU/dl)
* Currently on prophylactic therapy
* The same prophylaxis regimen in the last six months
* Age: 2 (with a body weight ≥12.5 kg ) - 45 years
* Adequate venous access
* Haemophilia patient's diary or equivalent regularly completed
* Ability of patient or family (for minors) to give informed consent
* Subject with health insurance

Exclusion Criteria:

* Age <2 and >45 years
* Haemophilia A with documented inhibitor in the last 12 months
* Clinically symptomatic liver disease (historical evidence documented in patient's medical file)
* Platelet count < 100x109/l
* Poor venous access
* Presence of a documented target joint
* Subject under legal protection measure.

Ages: 2 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-08-08 (Actual); Primary Completion 2019-09-08 (Estimated); Study Completion 2019-09-08 (Estimated)

PRIMARY OUTCOMES:
The correlation between the trough TGA (ETP) results of severe haemophilia patients who are on prophylaxis and the clinical efficacy of the ongoing prophylaxis regimen will be studied | The clinical efficacy of prophylaxis will be evaluated on the basis of the number of spontaneous joint bleeds the number of other relevant spontaneous bleeds and the consumption of clotting factor concentrate in the last 6 months prior to TGA.

SECONDARY OUTCOMES:
The correlation between the trough FVIII:C results of severe haemophilia patients who are on prophylaxis and the clinical efficacy of the ongoing prophylaxis regimen will be studied | The clinical efficacy of prophylaxis will be evaluated on the basis of the number of spontaneous joint bleeds the number of other relevant spontaneous bleeds and the consumption of clotting factor concentrate in the last 6 months prior to FVIII.

CONTACTS AND LOCATIONS:
Locations (7):
- France (7):
  - Hôpital Pellegrin, Bordeaux
  - Unité d'Hémostase Clinique Centre Régional de Traitement des Hémophiles Centre de Référence de Maladies Hémorragiques Hôpital Cardiologique Louis Pradel, Bron
  - CH Metropole Savoie site de Chambéry, Chambéry
  - CHU Dijon Bourgogne Hôpital François Mitterrand, Dijon
  - Chu Timone, Marseille
  - CHU de Nantes, Nantes
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne